CLINICAL TRIAL: NCT05838846
Title: Inhaled Versus Intravenous Milrinone for Patients Undergoing Mitral Valve Replacement Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed Ashraf Nasr, Assisstant Lecturer Anesthesia, Intensive care and Pain management - Faculty of Medicie - Menoufia University, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2/2023 ANET 60
Record Dates: First submitted 2023-04-06; First posted 2023-05-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Mitral Valve Replacement; Pulmonary Hypertension; Inhaled Milrinone; Intravenous Milrinone
Keywords: Milrinone; Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Milrinone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (iMil) (Experimental): Patients will receive 2 doses of inhaled milrinone at the following time points (after sternotomy and after aortic cross clamp off) at dosage of 50 mcg/kg by nebulization, inhaled milrinone will be administered through Aerogen solo with Pro-X controller - continuous mode- attached to ventilator circuit distal to viral/ bacterial heat and moisture exchange filter.
  Then pulmonary vascular resistance and systemic vascular resistance will be calculated after first dose ended by 2 minutes and after second dose ended by 15 minutes till stabilization of post CPB other variables like temperature and acid-base status, both measurements will be done while using inspired oxygen of 0.80.
  Interventions: Drug: Inhaled Milrinone
- Group B (IvMil) (Active Comparator): Patients will receive intravenous milrinone - started after induction of anesthesia - infusion at dosage of 0.3 - 0.75 mcg/kg/min after loading dose of 50 mic/kg over 10 min. After cross clamp off and temperature of 32 degree, Pulmonary vascular resistance and systemic vascular resistance will be calculated at the same corresponding time points to group A.
  Interventions: Drug: IV Milrinone

INTERVENTIONS:
Drug: Inhaled Milrinone — Patients will receive 2 doses of inhaled milrinone at the following time points (after sternotomy and after aortic cross clamp off) at dosage of 50 mcg/kg by nebulization, inhaled milrinone will be administered through Aerogen solo with Pro-X controller - continuous mode- attached to ventilator circuit distal to viral/ bacterial heat and moisture exchange filter.
  Arms: Group A (iMil)
Drug: IV Milrinone — Patients will receive intravenous milrinone infusion at dosage of 0.3 - 0.75 mcg/kg/min with loading dose of 50 mcg/kg over 10 min. After cross clamp off and temperature of 32 degree, Pulmonary vascular resistance and systemic vascular resistance will be calculated at the same corresponding time points to group A.
  Arms: Group B (IvMil)

SUMMARY:
This prospective open-label randomized study aims to compare the effect of inhaled versus intravenous milrinone on the pulmonary vascular resistance in patients undergoing mitral valve replacement surgery.

The primary outcome is to determine change in pulmonary artery pressure. The secondary outcomes include,

* Incidence of systemic hypotension.
* Hemodynamic affection and need of vasopressors and inotropes.
* Change in pulmonary vascular resistance versus systemic vascular resistance.
* Right ventricular function.
* Duration of mechanical ventilation.
* Need for mechanical circulatory support devices.
* Urine output
* Length of intensive care (ICU) in stay.

As the investigators hypothesize that inhaled milrinone has a selective pulmonary vasodilator effect devoid of the systemic hypotension with the intravenous administration.

DETAILED DESCRIPTION:
All patients underwent standard preoperative cardiac surgery assessment. Premedication included bromazepam and ranitidine, given the night before and 2 hours prior to arrival to OT. On arrival, IV access and arterial cannula were inserted under local anesthesia, along with routine monitoring electrocardiogram (ECG), pulse oximetery (SpO2), and IBP.

Anesthesia was induced with midazolam, fentanyl, and cis-atracurium. After tracheal intubation, ultrasound (US) guided- central venous catheter (CVC) was inserted and TEE also applied and then anesthesia maintained with morphine, cis-atracurium infusions, and sevoflurane. Mechanical ventilation was set to maintain end-tidal carbon dioxide (etco2) in the range of 30-40 mmHg using lung protective ventilation strategies.

During CPB, flow of 2.2 L.min-1.m-2, a custodiol cardioplegia was given, temperature kept at 28-32℃ and anesthesia maintained by sevoflurane- through a vaporizer mounted on CPB machine-.

A senior consultant certified cardiac anesthetist conducted a baseline TEE using Philips EPIQ CVxi echocardiography machine. Baseline measures included left ventricular ejection fraction (LVEF), and RV function represented by tricuspid annulus plane systolic excursion (TAPSE), fractional area changes (FAC), and right ventricular systolic pressure (RVSP) by doppler also, PVR and systemic vascular resistance (SVR) was calculated, plus patients hemodynamics (mean arterial blood pressure (MAP), heart rate (HR)), all measures were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Severe mitral regurgitation and moderate or severe pulmonary hypertension
* Scheduled for mitral valve replacement surgery

  # Criteria of severe mitral regurgitation:
* Central jet MR >40% LA or holosystolic eccentric jet MR
* Vena contracta ≥ 0.7 cm
* Regurgitant volume ≥60 ml
* Regurgitant fraction ≥50%
* EROA ≥0.40 cm2

  # Criteria of moderate and severe pulmonary hypertension:
* Moderate pulmonary hypertension; mean pulmonary artery pressure > 41 mmHg while, severe pulmonary hypertension; mean pulmonary artery pressure > 55 mmHg
* Mean pulmonary artery pressure > 40% of mean systemic blood pressure.
* Mean pulmonary artery pressure approximated from estimated systolic pulmonary artery pressure as following; mPAP= (estimated sPAP X 0.61) ± 2

Exclusion Criteria:

* Patients with aortic valvular lesions or pulmonary stenosis.
* Hemodynamic instability in the preoperative time (defined as acute requirement for vasoactive support or mechanical device).
* Contraindication to transesophageal echocardiography; esophageal stricture, tumor or diverticulum or active upper gastrointestinal bleeding
* Patients with hepatic or renal dysfunction.
* Patients with coagulopathy.
* Emergency surgeries.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary artery pressure | Intraoperative

SECONDARY OUTCOMES:
Incidence of systemic hypotension | Intraoperative
Hemodynamic affection and need of vasopressors and inotropes. | Intraoperative
Pulmonary vascular resistance versus systemic vascular resistance | Intraoperative
  Systemic vascular resistance: (MAP-CVP) x 80 / CO
  Pulmonary vascular resistance = (MPAP-PAWP) X 80 / CO
Right ventricular function | Intraoperative
  Measured by tricuspid annulus plane systolic excursion, fractional area changes, and right ventricular systolic pressure by doppler
Duration of mechanical ventilation | Postoperative in ICU (up to 24 hours)
Need for mechanical circulatory support devices | Intraoperative
Urine output | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Hassan, Professor, Study Chair — Faculty of Medicine - Menoufia University; Mohamed A Salem, A. Professor, Study Chair — Faculty of Medicine - Menoufia University; Khaled M Gaballah, A. Professor, Study Chair — Faculty of Medicine - Menoufia University; Mohammed O El Gouhary, Lecturer, Study Director — Faculty of Medicine - Ain Shams University
Locations (1):
- Menoufia University Hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No